CLINICAL TRIAL: NCT03143660
Title: Pediatric Practice-based Obesity Intervention to Support Families:FITLINE
Brief Title: FITLINE: Pediatric Practice-based Obesity Intervention to Support Families
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Responsible Party: Principal Investigator, Lori Pbert, Professor, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01HL130505 (NIH)
Record Dates: First submitted 2017-04-16; First posted 2017-05-08 (Actual); Last update posted 2022-01-31 (Actual); Status verified 2022-01

CONDITIONS: Obesity, Childhood
Keywords: obesity
MeSH Terms: conditions — Pediatric Obesity; Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Coaching (Active Comparator): A parent support component consisting of eight weekly telephone counseling calls by centrally located nutritionists to provide parents coaching tailored to their family's unique needs to help them set goals and make targeted lifestyle changes recommended by the American Academy of Pediatrics (AAP) for Stage 1, Prevention Plus, accompanied by a parent booklet
  Interventions: Behavioral: Coaching
- Materials (Active Comparator): Parents will receive the same educational materials provided in the Fitline family workbook mailed over 8 weeks to control for weekly contact and educational curriculum, but no Fitline counseling.
  Interventions: Behavioral: Materials

INTERVENTIONS:
Behavioral: Coaching — The eight weekly 30-minute Fitline calls provide personalized behavioral counseling and coaching to guide parents in improving their child's weight-related behaviors through targeted lifestyle changes recommended by the AAP for Stage 1, Prevention Plus. Calls are scheduled at a time convenient for the parent, including nights and weekends, with one nutritionist assigned to a family for consistency.
  Arms: Coaching
Behavioral: Materials — The workbook contains tips and practical strategies for implementing the AAP-recommended behavior changes discussed in the counseling sessions to support families in making lifestyle changes.
  Arms: Materials

SUMMARY:
The goal of this study is to investigate whether eight weekly telephone coaching sessions or materials on lifestyle interventions can be beneficial for overweight and obese 8-12 year olds.

DETAILED DESCRIPTION:
The proposed five-year cluster randomized controlled pediatric practice-based trial will compare the effectiveness of two practice-based interventions on improving diet and physical activity and reducing BMI among overweight and obese 8-12 year olds seen in pediatric practice: (1) Fitline-Coaching, consisting of a pediatric practice-based component plus Fitline counseling and workbook, or (2) Fitline-Workbook, consisting of the same practice-based component, but only the family workbook materials mailed over 8 weeks, with no referral to Fitline coaching. Sixteen pediatric primary care practices will be randomized to either the Fitline-Coaching (N=8) or the Fitline-Materials (N=8) condition. Five hundred and twelve parents and their children ages 8-12 with a body mass index (BMI) of > 85th percentile (overweight or obese) will be recruited from the practices to achieve N=400 at 12 month follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. child BMI >= 85th percentile for age/sex,
2. participating parent and child English speaking,
3. parent has access to a telephone and is available to participate in telephone counseling sessions, and
4. referred by the child's primary care provider.

Exclusion Criteria:

1. planning to move out of the area during the period of study participation,
2. medical condition that precludes adherence to AAP dietary and physical activity recommendations,
3. genetic or endocrine causes of obesity,
4. prescribed medications associated with weight gain,
5. child on psychiatric medications, and/or
6. morbidly obese (> 300 pounds). -

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 501 (Actual)
Dates: Start 2017-10-11 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-28 (Actual)

PRIMARY OUTCOMES:
Reducing BMI in overweight and obese children. | Baseline and 12-months post-baseline
  BMI will be calculated from weight (kg)/height squared (in meters) and BMI z-score for age/sex will be determined using CDC growth charts for the child. It is hypothesized that the Fitline-Coaching group compared to the Fitline-Workbook group will have greater reductions in BMI z-scores at 12-month follow-up
Reducing BMI in overweight and obese children. | Baseline and 6-months post-baseline
  BMI will be calculated from weight (kg)/height squared (in meters) and BMI z-score for age/sex will be determined using CDC growth charts for the child. It is hypothesized that the Fitline-Coaching group compared to the Fitline-Workbook group will have greater reductions in BMI z-scores at 6-month follow-up

SECONDARY OUTCOMES:
Improving the child's diet | Baseline and 6-months post-baseline
  It is hypothesized that the Fitline-Coaching group compared to the Fitline-Workbook group will have greater improvements in diet at 6-month follow-up. This will be measured by 24 hour dietary recalls conducted 3 times at each time point.
Improving the child's diet | Baseline and 12-months post-baseline
  It is hypothesized that the Fitline-Coaching group compared to the Fitline-Workbook group will have greater improvements in diet at 12-month follow-up. This will be measured by 24 hour dietary diet recalls conducted three times at each time point.
Improving the child's physical activity | Baseline and 6-months post-baseline
  It is hypothesized that the Fitline-Coaching group compared to the Fitline-Workbook group will have greater improvements in their level of physical activity at 6-month follow-up. This will be measured by the Physical Activity Questionnaire (PAQ-C).
Improving the child's physical activity | Baseline and 12-months post-baseline
  It is hypothesized that the Fitline-Coaching group compared to the Fitline-Workbook group will have greater improvements in their level of physical activity at 12-month follow-up. This will be measured by the Physical Activity Questionnaire (PAQ-C).
Effect of the Fitline-Coaching on BMI through a composite measure of Social Cognitive Theory constructs | Baseline and 6-months post-baseline
  It is hypothesized that the effect of the Fitline-Coaching on child BMI will be predicted by changes in Social Cognitive Theory constructs. Parents will complete a survey assessing: (1) anticipated benefits of the behavior change (outcome expectations) (23-item questionnaire); (2) perceived support and barriers to addressing their child's behavior changes (15-item questionnaire); (3) self efficacy in helping their child improve their diet and physical activity (12-item) questionnaire; (4) behavioral capability (12-item questionnaire); and (5) knowledge (7-item questionnaire).
  Children will complete a survey assessing (1) anticipated benefits of the behavior change (outcome expectations) (23-item questionnaire); (2) perceived support and barriers (67-item questionnaire); (3) self efficacy (16-item questionnaire); (4) behavioral capability (12-item questionnaire); and (5) knowledge (7 item questionnaire).
Effect of the Fitline-Coaching on BMI through a composite measure of Social Cognitive Theory constructs | Baseline and 12-months post-baseline
  The effect of the Fitline-Coaching on child BMI will be predicted by changes in Social Cognitive Theory constructs. Parents will complete a survey assessing: (1) the anticipated benefits of the behavior change (outcome expectations) using a 23-item questionnaire; (2) parent's perceived support and barriers to addressing their child's behavior changes using a 15 item questionnaire; (3) parent's self efficacy in helping their child improve their diet and physical activity using a 12 item questionnaire; (4) behavioral capability using a 12 item questionnaire; and (5) knowledge utilizing a 7 item questionnaire.
  Children will complete a survey assessing (1) the anticipated benefits of the behavior change (outcome expectations) using a 23-item questionnaire; (2) their perceived support and barriers a 67-item questionnaire; (3) child's self efficacy using a 16-item questionnaire; (4) behavioral capability using a 12-item questionnaire; and (5) knowledge utilizing a 7-item questionnaire.
Cost Effectiveness | Baseline and 12-months post-baseline
  Costs and health outcomes will be compared across conditions. Costs will include those of: (1) provider training and intervention, (2) office set-up and support, (3) intervention materials, and (4) Fitline coaching. The outcome will be change in BMI z-score.
Cost Effectiveness | Baseline and 12-months post-baseline
  Costs and health outcomes will be compared across conditions. Costs will include those of: (1) provider training and intervention, (2) office set-up and support, (3) intervention materials, and (4) Fitline coaching. The outcome will be change in quality of life as measured by the quality adjusted Pediatric Quality of Life Inventory (PedsQL 4.0) scores.

CONTACTS AND LOCATIONS:
Overall Officials: Lori Pbert, PhD, Principal Investigator — University of Massachusetts, Worcester
Locations (1):
- University of Massachusetts, Worcester, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pbert L, Trivedi M, Druker S, Bram J, Olendzki B, Crawford S, Frisard C, Andersen V, Waring ME, Clements K, Schneider K, Geller AC. Supporting families of children with overweight and obesity to live healthy lifestyles: Design and rationale for the Fitline cluster randomized controlled pediatric practice-based trial. Contemp Clin Trials. 2021 May;104:106348. doi: 10.1016/j.cct.2021.106348. Epub 2021 Mar 8. PMID 33706002